CLINICAL TRIAL: NCT03210883
Title: Global Electrical Heterogeneity and Clinical Outcomes
Acronym: GEHCO
Status: Completed | Type: Observational
Sponsor: Larisa Tereshchenko (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Larisa Tereshchenko, Associate Professor of Medicine, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Other Study IDs: STUDY00016754
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure; Implantable Defibrillator User; Ventricular Arrythmia
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective multicenter cohort will validate an independent association of electrocardiographic (ECG) global electrical heterogeneity (GEH) measures with sustained ventricular tachyarrhythmias and appropriate ICD therapies in systolic heart failure patients with primary prevention ICD, and will validate and re-calibrate GEH ECG risk score for prediction of sustained ventricular tachyarrhythmias and appropriate ICD therapies in systolic heart failure patients with primary prevention ICD.

ELIGIBILITY:
Inclusion Criteria:

* records of systolic heart failure patients with primary prevention ICDs/CRT-Ds implanted for routine clinical indications

Exclusion Criteria:

* absent baseline pre-implant digital ECG;
* missing data on clinical predictors and covariates;
* missing ICD programming data (including number of intervals to detect [NID] or time to detect, number of detection zones, heart rate for each detection zone, and anti-tachycardia pacing [ATP] programming);
* missing outcomes data.
* records of patients with inherited channelopathies (e.g. long QT syndrome, Brugada syndrome), inherited cardiomyopathies (e.g. hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy), and congenital heart disease.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective records of systolic heart failure patients with primary prevention ICDs/CRT-Ds implanted for routine clinical indications
Sampling Method: Probability Sample
Enrollment: 3471 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome: sustained VT/VF event with appropriate ICD therapy (either ATP or shock) | up to 15 years
  Sustained ventricular tachyarrhythmia event with appropriate ICD therapy (either antitachycardia pacing or shock)
Primary competing outcome: All-cause death without preceding sustained VT/VF with appropriate ICD therapy | up to 15 years
  All-cause death without preceding sustained ventricular tachyarrhythmia with appropriate ICD therapy

SECONDARY OUTCOMES:
sustained monomorphic ventricular tachycardia | up to 15 years
  Sustained monomorphic ventricular tachycardia with appropriate ICD therapies (either antitachycardia pacing or ICD shock)
sustained polymorphic ventricular tachycardia / ventricular fibrillation | up to 15 years
  sustained polymorphic ventricular tachycardia or ventricular fibrillation with appropriate ICD therapies (either antitachycardia pacing or ICD shock)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa G Tereshchenko, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oregon Health and Science University, Portland, Oregon
  - Veteran Administration Portland Healthcare System, Portland, Oregon

REFERENCES:
- [Background] Waks JW, Hamilton C, Das S, Ehdaie A, Minnier J, Narayan S, Niebauer M, Raitt M, Tompkins C, Varma N, Chugh S, Tereshchenko LG. Improving sudden cardiac death risk stratification by evaluating electrocardiographic measures of global electrical heterogeneity and clinical outcomes among patients with implantable cardioverter-defibrillators: rationale and design for a retrospective, multicenter, cohort study. J Interv Card Electrophysiol. 2018 Jun;52(1):77-89. doi: 10.1007/s10840-018-0342-2. Epub 2018 Mar 14. PMID 29541969
- [Result] Waks JW, Haq KT, Tompkins C, Rogers AJ, Ehdaie A, Bender A, Minnier J, Dalouk K, Howell S, Peiris A, Raitt M, Narayan SM, Chugh SS, Tereshchenko LG. Competing risks in patients with primary prevention implantable cardioverter-defibrillators: Global Electrical Heterogeneity and Clinical Outcomes study. Heart Rhythm. 2021 Jun;18(6):977-986. doi: 10.1016/j.hrthm.2021.03.006. Epub 2021 Mar 6. PMID 33684549
- [Result] Haq KT, Javadekar N, Tereshchenko LG. Detection and removal of pacing artifacts prior to automated analysis of 12-lead ECG. Comput Biol Med. 2021 Jun;133:104396. doi: 10.1016/j.compbiomed.2021.104396. Epub 2021 Apr 19. PMID 33872969
- [Derived] Tereshchenko LG, Waks JW, Tompkins C, Rogers AJ, Ehdaie A, Henrikson CA, Dalouk K, Raitt M, Kewalramani S, Kattan MW, Santangeli P, Wilkoff BW, Kapadia SR, Narayan SM, Chugh SS. Competing risks of monomorphic vs. non-monomorphic ventricular arrhythmias in primary prevention implantable cardioverter-defibrillator recipients: Global Electrical Heterogeneity and Clinical Outcomes (GEHCO) study. Europace. 2024 Jun 3;26(6):euae127. doi: 10.1093/europace/euae127. PMID 38703375